CLINICAL TRIAL: NCT00467844
Title: Double-Blind, Placebo-Controlled, Dose-Finding Study of the Effect of GTx-024 on Muscle Wasting (Cachexia) in Patients With Cancer
Brief Title: Study of GTx-024 on Muscle Wasting (Cachexia) Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: G200502; NCT00832104 (obsolete NCT alias)
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Cachexia
Keywords: Cachexia; Muscle Wasting; Non-Small Cell Lung Cancer; Colorectal Cancer; Non-Hodgkin's Lymphoma; Stage 3 or 4 Breast Cancer; Chronis Lymphocytic Leukemia
MeSH Terms: conditions — Cachexia; Muscular Atrophy; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lymphoma, Non-Hodgkin | interventions — ostarine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 1 mg GTx-024
  Interventions: Drug: GTx-024
- 2 (Experimental): 3 mg GTx-024
  Interventions: Drug: GTx-024
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GTx-024 — 1 mg GTx 024
  Arms: 1
Drug: GTx-024 — 3 mg GTx-024
  Arms: 2
Drug: Placebo — Matching Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to assess if Gtx-024 is effective in increasing lean body mass in subjects with muscle wasting related to cancer.

DETAILED DESCRIPTION:
Cancer cachexia is characterized by a hypermetabolic state that leads to catabolism that is responsible for reductions in lean mass.These catabolic changes are accompanied by an increase in total energy expenditure, but a decrease in voluntary energy expenditure that ultimately results clinically in cachexia and its symptoms of lethargy, fatigue, weakness and general malaise (Kotler DP. Cachexia. Ann Intern Med. 2000; 133:622-634).

The prevalence of cachexia increases from 50 percent at presentation to more than 80 percent before death from malignancy. In over 20 percent of cancer patients, cachexia is the cause of death (Bruera E. Anorexia, cachexia and nutrition. Br Med J 1997;315:1219-1222). Cancer cachexia leads to shorter survival, decreased response rates and increased toxicity to chemotherapy, weakness, and an overall decreased quality of life (DeWys et al. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7). The purpose of this study is to assess the efficacy of GTx-024 on total body lean mass. Secondary endpoints include but are not limited to assessment of GTx-024 on muscle function, total body weight and total body fat mass.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, subjects must meet all of the following criteria:

* have been diagnosed with Stage 2, 3 or 4 non-small cell lung cancer or Stage 2, 3 or 4 colorectal cancer or non-hodgkin's lymphoma or chronic lymphocytic leukemia or Stage 3 or 4 breast cancer.
* be prior to initiation of or between cycles of chemotherapy.
* have experienced greater than or equal to 2% weight loss from the highest patient reported weight in the 6 months prior to screening for Protocol G200502 (Wt = body weight)

  % weight loss = (Wt at screening - highest Wt in last 6 months) / highest Wt in last 6 months x 100%
* If surgery is part of the cancer treatment, screening for this study should be conducted at least 2 weeks (14 days) after surgery.
* have a life expectancy of >6 months
* FEMALES - be clinically confirmed as postmenopausal
* MALES - over 45 years of age
* ECOG score ≤1

Exclusion Criteria:

Subjects with any of the following will NOT be eligible for enrollment in this study:

* history of active/uncontrolled congestive heart failure, chronic hepatitis, hepatic cirrhosis, or HIV infection
* Cardiovascular: No uncontrolled hypertension
* Positive screen for Hepatitis B consisting of HBsAg (Hepatitis B Surface Antigen), anti-HCV (Hepatitis C Antibody), hepatitis A antibody IgM, or HIV
* Currently taking testosterone, OXANDRIN® (oxandrolone), testosterone-like agents (such as DHEA, androstenedione, and other androgenic compounds, including herbals), or antiandrogens (Please note that previous therapy with testosterone and testosterone-like agents is acceptable with a 30 day wash-out. However, if the previous testosterone therapy was a long-term depot, within the past 6 months, the site should call the medical monitor for this study to determine appropriate washout period.)
* Currently taking megestrol acetate (MEGACE®), dronabinol (MARINOL®), or any prescription medication intended to increase appetite or treat unintentional weight loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (49):
  - Alaska Cancer Research and Education Center, Anchorage, Alaska
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Compassionate Cancer Care, Corona, California
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Compassionate Cancer Care, Riverside, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Dorcy Cancer Center, Pueblo, Colorado
  - Hartford Hospital Cancer Clinical Research Office, Hartford, Connecticut
  - Medical Oncology & Hematology, PC, Waterbury, Connecticut
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - The Radiation Oncology Group, Lake Worth, Florida
  - Watson Clinic LLP, Center for Cancer Care & Research, Lakeland, Florida
  - Osler Medical, Melbourne, Florida
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - Dublin Hematology and Oncology, Dublin, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Johns Hopkins University Clinical Trial Unit, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - The Center for Clinical Research WA County Hospital, Hagerstown, Maryland
  - Newland Medical Center, Southfield, Michigan
  - The West Clinic, Corinth, Mississippi
  - West Clinic, Corinth, Mississippi
  - The West Clinic, Southaven, Mississippi
  - West Clinic, Southaven, Mississippi
  - Hematology & Oncology Associates at Bridgeport, Tupelo, Mississippi
  - Heartland Hematology-Oncology Associates, Kansas City, Missouri
  - Donald H. Berdeaux, MD, FACP, PC, Great Falls, Montana
  - Great Falls Clinic, LLP - Clinic Cancer Care, Great Falls, Montana
  - Creighton University Hematology/Oncology Clinic, Omaha, Nebraska
  - Cancer Care of Western North Carolina, Ashville, North Carolina
  - Four Seasons Hospice & Palliative Care, Flat Rock, North Carolina
  - Hanover Medical Specialists, Wilmington, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Hematology Oncology Consultants, Worthington, Ohio
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Berks Hematology-Oncology Associates, West Reading, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - West Clinic, Memphis, Tennessee
  - Dallas Oncology Consultants, Dallas, Texas
  - Providence Everett Medical Center, Cancer Research Department, Everett, Washington
- Canada (2):
  - University of Alberta Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Dobs AS, Boccia RV, Croot CC, Gabrail NY, Dalton JT, Hancock ML, Johnston MA, Steiner MS. Effects of enobosarm on muscle wasting and physical function in patients with cancer: a double-blind, randomised controlled phase 2 trial. Lancet Oncol. 2013 Apr;14(4):335-45. doi: 10.1016/S1470-2045(13)70055-X. Epub 2013 Mar 14. PMID 23499390

RESULTS

PARTICIPANT FLOW:
Groups:
- GTx -024: 1 mg
- GTx-024: 3 mg
- 3 mg of Placebo: Placebo
Period: Overall Study
Arm/Group | GTx -024 | GTx-024 | 3 mg of Placebo
Started | 53 | 54 | 52
Completed | 34 | 34 | 38
Not Completed | 19 | 20 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GTx -024 | GTx-024 | 3 mg of Placebo | Total
Number analyzed (Participants) | 53 | 54 | 52 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 24 | 71
  >=65 years | 28 | 32 | 28 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (10.03) | 66.3 (10.51) | 65.6 (8.73) | 65.9 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 17 | 56
  Male | 34 | 34 | 35 | 103
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 36 | 112
  Argentina | 14 | 17 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of GTx-024 on Total Body Lean Mass.
Description: Change in total body lean mass as measured by dual energy x-ray absorptiometry (DEXA)from baseline to 4 months.
Time Frame: Baseline to Four Months
Population: The number of participants were those subjects in the modified intent-to-treat population (defined as subjects with at least one post baseline DEXA for LBM) who had baseline and 4 month DEXA results for LBM (observed cases).
Measure: Median (Full Range); unit: kg
Groups:
- Placebo: Placebo
Arm/Group | GTx-024 1 mg | GTx-024 3 mg | Placebo
Number analyzed (Participants) | 32 | 34 | 34
kg | 1.55 [-2.06 to 12.64] | 0.98 [-4.84 to 11.54] | 0.02 [-5.81 to 7.46]

2. Secondary Outcome: To Assess the Efficacy of GTx-024 on Muscle Function (Performance) as Measured by Stair Climb.
Description: Change in stair climb power from baseline to 4 months. Stair climb power is defined power (watts)=[9.8 m/sec**2]*[weight (kg)]*[height of 12 steps(meters)]/ [time (seconds) up the 12 steps].
Time Frame: Four Months
Population: The subjects were in the MITT population (had a post baseline DEXA) and had a month 4 stair climb assessment (observed cases).
Measure: Median (Full Range); unit: watts
Arm/Group | GTx -024 | GTx-024 | 3 mg of Placebo
Number analyzed (Participants) | 31 | 28 | 36
watts | 19.93 [-235.3 to 110.1] | 12.84 [-77.7 to 93.1] | 11.34 [-156.4 to 56.4]

ADVERSE EVENTS:
Arm/Group | GTx -024 | GTx-024 | 3 mg of Placebo
Serious Adverse Events (participants affected / at risk) | 14/53 | 15/54 | 17/52
Other Adverse Events (participants affected / at risk) | 47/53 | 49/54 | 46/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GTx -024 (N=53) | GTx-024 (N=54) | 3 mg of Placebo (N=52)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 0 (0) | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
rectal obstruction (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 1 | 0 (0)
diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1
pneumonia (Infections and infestations) | 2 | 3 | 2
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1
septic shock (Infections and infestations) | 0 (0) | 1 | 0 (0)
staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1
compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
patella fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 1
road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0/0 (0) | 1 (1)
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 7 | 8 (9)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 | 0 (0)
metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 | 0 (0)
non small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx -024 (N=53) | GTx-024 (N=54) | 3 mg of Placebo (N=52)
anaemia (Blood and lymphatic system disorders) | 13 | 7 | 8
neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 2
thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 3
abdominal pain (Gastrointestinal disorders) | 2 | 8 | 3
constipation (Gastrointestinal disorders) | 9 | 6 | 2
diarrhoea (Gastrointestinal disorders) | 8 | 9 | 7
vomiting (Gastrointestinal disorders) | 9 | 4 | 6
asthenia (Gastrointestinal disorders) | 1 | 7 | 4
fatigue (Gastrointestinal disorders) | 8 | 14 | 11
pyrexia (General disorders) | 5 | 8 | 3
pneumonia (Infections and infestations) | 2 | 4 | 2
weight decreased (Investigations) | 5 | 8 | 5
anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 | 2 (2)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 6 (6)
back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (4)
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 8 (8) | 8 (9)
headache (Nervous system disorders) | 3 (3) | 5 (7) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) | 6 (6)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 13 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less